CLINICAL TRIAL: NCT00272077
Title: Pilot Study on Glycaemic Variability in Type 2 Diabetes Mellitus Patients With Basal Insulin and Fixed Combo Oral Antidiabetic Treatment.
Brief Title: Insulin Glargine in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_3509; EudraCT # : 2004-002730-19
Record Dates: First submitted 2006-01-02; First posted 2006-01-04 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: Insuline glargine

SUMMARY:
Primary objective:

To evaluate in explorative manner the fasting blood glucose (FBG) coefficient of variability (CV)calculated on SMBG values (SMBG : Self-Monitoring of Blood Glucose).

Secondary objectives:

The secondary objectives are the assessment of: changes in glycaemic control (HbA1C), frequency of hypoglycaemias, changes in weight, final insulin dose, changes in lipid parameters, changes in urinary albumin-to-creatinine ratio, profile of patient which best fits each of the algorithms with the dependent variable of change in HbA1C and independent variables of age, gender, race, tobacco use, diabetes complications, initial HbA1C, initial weight, duration of diabetes mellitus, general education and diabetes education.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus for at least 5 years;
* Treatment with oral antidiabetic drugs in fixed combination (Combo, i.e. glibenclamide 2.5 mg + metformin 400 mg, 2 or 3 tablets, at stable dose in the last 3 months);
* HbA1c >= 8% and <= 11%;
* Body mass index (BMI) > 27 and < 35 kg/m2;
* Willingness and demonstrated ability to inject insulin;
* Demonstrated ability and willingness to perform self-monitoring of blood glucose (SMBG);

Exclusion criteria:

* Patients diagnosed with type 1 insulin dependent diabetes;
* Patients with latent autoimmune diabetes of adults (LADA), defined as fasting C-peptide levels < 1 ng/ml;
* Cardiac status NYHA III-IV;
* Impaired renal function as shown by (but not limited to) serum creatinine >= 1.5 mg/dl for males or >= 1.4 mg/dl for females;
* Planned pregnancy, pregnant or lactating females;
* Failure to use adequate contraception (women of current reproductive potential only);
* Any current malignancy, previous breast cancer, or malignant melanoma within the past 5 years;
* Diagnosis of dementia
* Hypersensitivity to insulin or any of their components or to metformin;
* Current or previous insulin therapy other than during hospitalisations;
* Inability or unwillingness to continue metformin at study dosages throughout the study;
* Treatment with intermittent doses of systemic steroids or large doses of inhaled steroids for the past one year (fixed doses for the past 6 months is acceptable providing there is no plan to change the dosage regime);
* Stroke, Myocardial Infarction (MI), Coronary Artery Bypass Graft (CABG), Percutaneous Transluminal Coronary Angioplasty (PTCA), or Angina Pectoris within the last 12 months;
* History of drug or alcohol abuse;
* Receipt of an experimental drug or use of an experimental device within the 30 days prior to study entry;

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-04; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
SMBG values | during the last 4 weeks before visit 3 (end of cycle 1) and visit 4

SECONDARY OUTCOMES:
glycaemic control (HbA1c, fasting blood glucose, insulin and C-peptide), | During the study conduct
frequency of hypoglycaemias | During the study conduct
body weight | During the study conduct
final insulin dose | During the study conduct
lipid profile (serum total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides) | During the study conduct
urinary albumin-to-creatinine ratio | During the study conduct
standard meal test | during the study conduct
results of CGMS | During the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: PAIZIS GEORGES, MD, Study Director — Sanofi